CLINICAL TRIAL: NCT02723461
Title: Randomised Controlled Trial Comparing Continuous Intravenous Oxytocin Infusion With Pulsatile Administration of Intravenous Oxytocin for Augmentation of the First Stage of Labor
Brief Title: Continuous Oxytocin Infusion Versus Pulsatile Intravenous Oxytocin for Augmentation of First Stage of Labor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pulsatile oxytocin
Record Dates: First submitted 2016-03-26; First posted 2016-03-30 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Failed Induction (of Labor) by Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulsatile oxytocin (Active Comparator): Using a programmable syringe pump, the pulsatile regime, oxytocin (Syntocinon, stock solution: 10 iU/mL) will be administered for 10 seconds every 6 minutes and the dose (2 mU/pulse) doubled every 30 minutes until uterine contractions will be established (3-4 in 10 minutes). This regime stems from the observation that physiologic oxytocin may be released in a pulsatile fashion every 4-6 minutes (Dawood et al.,1979)
  Interventions: Drug: Pulsatile Oxytocin
- continuous oxytocin (Active Comparator): Continuous group will be administrated oxytocin (Syntocinon, stock solution: 10 iU/mL) at starting dose (2 mU/min) in a continuous manner doubled every 30 minutes until uterine contractions will be established (3-4 in 10 minutes).
  Interventions: Drug: Continuous Oxytocin

INTERVENTIONS:
Drug: Pulsatile Oxytocin — Using a programmable syringe pump, oxytocin will be administered for 10 seconds every 6 minutes and the dose (2 mU/pulse) doubled every 30 minutes until uterine contractions will be established (3-4 in 10 minutes).
  Other Names: syntocinon
  Arms: pulsatile oxytocin
Drug: Continuous Oxytocin — Oxytocin will be administered at starting dose (2 mU/min) in a continuous manner doubled every 30 minutes until uterine contractions will be established (3-4 in 10 minutes).
  Other Names: syntocinon
  Arms: continuous oxytocin

SUMMARY:
Comparing continuous intravenous oxytocin infusion with pulsatile administration of intravenous oxytocin for augmentation of the first stage of labor.

DETAILED DESCRIPTION:
The study population comprises120 cases with spontaneous onset of labor who are admitted to the labor ward at causalities of Ain shams university maternity hospital.

The required sample size has been calculated using the IBM© SamplePower© Software (IBM© Corp., Armonk, NY, USA). A previous study by Tribe et al., 2012 reported that the mean infusion to delivery time associated with continuous infusion of oxytocin was 7.17 hours with a 95% confidence interval (95% CI) of 6.58 to 7.77 hours versus 9.61 hours (95% CI, 8.95 to 10.27 hours) in association with pulsatile oxytocin. The sample size for either regimen in that study was 240 patients or 241 patients, respectively. From the study of Tribe et al. (2012), it could be estimated that the standard deviation (SD) for the infusion to delivery time was 4.66 hours or 5.23 hours for the continuous or pulsatile oxytocin regimen, respectively. This calculation is derived from solving any of the following equations for the SD given the mean, lower or upper 95% CI limit, and sample size:

Lower 95% CI limit = mean - (1.96 * SD / √n)..... Equation 1 Upper 95% CI limit = mean + (1.96 * SD / √n…..Equation 2 where SD is the standard deviation and n is the sample size (Chow et al., 2003).

So, it is estimated that a sample size of 66 patients in either study group (total, 132 patients) would achieve a power of 80% (type II error, 0.2) to detect a statistically significant difference between the two groups as regards the infusion to delivery time using a two-side unpaired Student t test with a confidence level of 95% (type I error, 0.05). the mean ± SD infusion to delivery time in both groups is assumed to be identical and to equal 9.61 ± 5.23 hours under the null hypothesis. Under the alternative hypothesis, the mean ± SD infusion to delivery time is assumed to equal 7.17 ± 4.66 hours in the continuous infusion group versus 9.61 ± 5.23 hours in the pulsatile group.

This sample size of 66 patients in each study group would have a power of 93% (type II error, 0.07) to detect a statistically significant difference between the two groups as regards the rate of successful induction of labor for a medium effect size (w) of 0.3 using a two-sided chi-squared test with a confidence level of 95% (type I error, 0.05). The effect size (w) is calculated as follows:

w =√(χ^2/N), where χ2 is the chi-squared statistic and N is the total sample size. (Chow et al., 2003).

Following admission, all patients will undergo complete clinical examination and detailed medical history will be obtained as follows:

A. Personal history. B. Obstetric history: where the gestational age will be calculated by the date of last menstrual period or by ultrasonography in unreliable dates.

C. Gynecological history.

Grouping:

The patients needing augmentation of first stage of labor will be divided equally into two groups:

Group 1 (study group ; 60 patients ) :

Patients at labor are given augmentation by oxytocin in pulsatile method

Group 2 (control group ;60 patients) :

Patients at labor are given augmentation by oxytocin in continuous method

Intervention:

Pulsatile group:

Pulsatile infusion protocol using a programmable syringe pump is applied .The pulsatile regime, oxytocin (Syntocinon,stock solution: 10 iU/mL) will be administered for 10 seconds every 6 minutes and the dose (2 mU/pulse) will be doubled every 30 minutes until uterine contractions will be established (3-4 in 10 minutes). This regime stems from the observation that physiologic oxytocin may be released in a pulsatile fashion every 4-6 minutes (Dawood et al.,1979)

Continuous group :

Continuous group will be administrated oxytocin (Syntocinon,stock solution: 10 iU/mL) at starting dose (2 mU/min) in a continuous manner doubled every 30 minutes until uterine contractions will be established (3-4 in 10minutes).

Then each patient will have case record form in which the following data will be recorded:

1. Patient initials.
2. Study number.
3. Group.
4. Parity.
5. Gestatinal age ( first day of last menstrual period - early ultrasound).
6. Rupture of membranes.
7. Duration of rupture of membranes.
8. Duration of first stage of labour.
9. Duration of second stage of labour.
10. Need for instrumental delivery.
11. Need for Cesarean section.
12. Adverse effect.
13. Neonatal outcome.
14. Maternal complications.
15. Adverse effect related to oxytocin.
16. Total dose of oxytocin infused.
17. Previous complicated vaginal delivery.

ELIGIBILITY:
Inclusion Criteria

1. Women in labor (cervical dilatation 3-4 centimeters) who require augmentation of first stage of labor.
2. Single viable fetus.
3. Rupture of membranes before augmentation of labor.
4. Cephalic presentation.
5. Term pregnancy.

Exclusion Criteria:

1. Malpresentation.
2. Induction of labor by prostaglandins.
3. Any uterine previous surgery.
4. Fetal anomalies.
5. Premature labor.
6. Previous cesarean section.
7. Any uterine anomalies.
8. Multiple pregnancy.

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
duration of active phase of first stage of labor | 24 hours
  The time in hours from start of infusion of pulsatile oxytocin at onset of established labor (cervical dilatation 3-4 cm ) to the end of first stage of labour (cervical dilatation 10 cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided